CLINICAL TRIAL: NCT06824675
Title: Point-of-care Ultrasound Teledidactic Teaching for Prehospital Emergency Personnel
Acronym: POCUS TT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Semmelweis University Budapest (Unknown); Ludwig Boltzmann Institute Digital Health and Patient Safety (Other)
Responsible Party: Principal Investigator, Josef Michael Lintschinger, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2107/2024
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-02

CONDITIONS: eFast; Fate; Education, Medical; Point of Care Ultrasound (POCUS)
Keywords: EMS Personell; Education; Medical Education; critical care; emergency; Ultrasound; POCUS; Anaesthesiology; emergency medical technician; point-of-care ultrasound
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: The study consists of five phases. Participants begin by watching an introductory video and completing an electronic questionnaire to provide baseline information, including prior POCUS experience and openness to new methods. They are then randomly assigned to either the teledidactic (intervention) or in-person (control) training group.
  Next, all participants complete a standardized e-learning course covering POCUS basics and the eFAST protocol. This is followed by a supervised hands-on training session conducted either in person or remotely, based on group assignment.
  Participants are then evaluated during a simulated emergency case. They also complete a follow-up questionnaire on their cognitive load and learning experience.
  Finally, expert reviewers analyze video recordings of the assessments using the OSAUS scoring system to evaluate systematic examination skills and image interpretation accuracy
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Teledidactic Training (Other): Remote, online hands-on training
  Interventions: Other: Teledidactic Training
- In-Person Hands-on Training (Other): Traditional face-to-face hands on-training
  Interventions: Other: In-Person Hands-on Training

INTERVENTIONS:
Other: Teledidactic Training — Participants will take part in a tele-didactic training session, matching the duration of the control group's training. This workshop will cover the same content as the control group's session, but instead of in-person instruction, teaching experts will deliver the training remotely using telemedicine software.
  Arms: Teledidactic Training
Other: In-Person Hands-on Training — Participants will attend a face-to-face, hands-on workshop led by experts to learn the eFAST protocol.
  Arms: In-Person Hands-on Training

SUMMARY:
The goal of this clinical trial is to compare two methods of teaching emergency medical service (EMS) providers how to use point-of-care ultrasound (POCUS) to quickly assess critical conditions like internal bleedings. The main questions it aims to answer are:

Is teledidactic training as effective as face-to-face training in teaching POCUS skills? What are the participants' experiences, cognitive load, and feedback regarding these training methods? Researchers will compare remote, online hands-on training (teledidactic training) to traditional, face-to-face hands-on training (in-person training) to see if remote training is equally effective.

Participants will:

Be EMS providers from Austria and Hungary, aged 18 years or older, with no extensive prior experience in POCUS.

Be randomly assigned to either the tele-didactic or in-person training group (50 participants per group).

Undergo training sessions designed to teach POCUS skills and provide feedback on their learning experience.

This study is part of the European Union-funded Digi4Care project, which aims to promote digitalization in healthcare. It is significant because, if remote training proves effective, it could provide high-quality education to EMS providers in rural or underserved areas, ensuring they have the necessary skills to assess and respond to critical conditions.

DETAILED DESCRIPTION:
POCUS is a valuable tool that helps EMS providers quickly assess critical conditions like internal bleeding or heart problems, which can be crucial in emergency situations. However, many rural and remote areas with limited infrastructure face challenges, such as restricted access to hands-on training and specialized instructors. This study aims to compare two educational approaches - teledidactic versus traditional in-person hands-on training - for teaching EMS providers the skills necessary to perform POCUS based on the eFAST protocol.

In this study participants will be devided into the intervention group (teledidactic training) and the control group (in-person training)

1. Teledidactic Training: This involves remote, online hands-on training.
2. In-Person Training: This is the traditional face-to-face hands-on training. Participants in this study are EMS providers from Austria and Hungary who are at least 18 years old and do not have extensive prior experience with POCUS. A total of 100 participants will be randomly assigned to either the teledidactic or in-person training group.

The primary objective of the study is to compare the effectiveness of teledidactic versus in-person training in teaching POCUS skills. Secondary objectives include evaluating participants' experiences with these teaching methods, their cognitive load during the learning process, and their feedback on the training methods.

This study is important because it seeks to determine if remote training can be as effective as in-person training. If successful, this could help provide high-quality education to EMS providers in rural or underserved areas, ensuring they have the necessary skills to quickly assess and respond to critical conditions. The study is part of the European Union-funded Digi4Care project, which aims to promote digitalization in healthcare.

All collected data will be securely stored and anonymized to protect participants' privacy. The study follows ethical guidelines to ensure participants' rights and safety. Participation is voluntary, and participants can withdraw at any time.

ELIGIBILITY:
Inclusion Criteria:

* EMT-Intermediate/Advanced in the Austrian or Hungarian EMS
* ≥18 years

Exclusion Criteria:

* Experienced POCUS examiners, defined as >20 real-life or simulated POCUS examinations following the eFAST protocol
* inadequate knowledge of English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-02-23 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Difference in the performance of an eFAST POCUS examination between randomized groups | evaluation within 3 weeks after study completion
  The primary outcome measure is the difference in the total Objective Structured Assessment of Ultrasound Skill (OSAUS) score between the participants' of the two groups. Possible assessment scores range from 7 to 37 points, with higher scores indicating better performance.

SECONDARY OUTCOMES:
Difference in OSAUS score for each objective between randomized groups | evaluation within 3 weeks after study completion
  The evaluation of different objectives within the two intervention groups using the respective OSAUS score for each individual objective. Objectives: indication for the examination; applied knowledge of ultrasound equipment; image optimization; systematic examination, interpretation of images, documentation of examination, medical decision making.
Difference in time taken to demonstrate all views as required by the assessment checklist | evaluation within 3 weeks after study completion
  Evaluation of the time taken to demonstrate all required views listed on the checklist. Views: Right Upper Quadrant (Subphrenic space, right costodiaphragmatic recess, hepatorenal space, liver, right kidney); Left Upper Quadrant (Subphrenic space, left costodiaphragmatic recess, splenorenal recess, spleen, left kidney); Pelvic view (rectouterine such in females or rectovesical such in males); Cardiac View subcostal (4-chamber view); Lungs (left and right) (pleural sliding including M-Mode image, Presence or absence of B-Lines)
Difference in cognitive load between randomized groups | evaluation within 3 weeks after study completion
  Assessment of the cognitive load using the NASA Task load index for overall cognitive load and for each individual objective (mental demand, physical demand, temporal demand, performance, effort, frustration)
Difference in learning outcomes and training design using TEI between randomized groups | evaluation within 3 weeks after study completion
  Compare learning outcomes and training design between randomized groups using the Training Evaluation Inventory (TEI). Learning outcomes include subjective fun, perceived usefulness, difficulty, knowledge growth, and attitudes toward the training. Training design elements such as problem-based learning, activation of prior knowledge, demonstration, application, and integration will also be assessed. These aspects will be measured with a 45-item inventory using a 5-point Likert scale, ranging from "I do not agree" to "I agree very much," providing insights into the effectiveness of the training methods.
Evaluation of participants' feedback on specific questions | evaluation within 3 weeks after study completion
  Evaluation of participants' feedback on their learning experience using specific questions. Participants will rate, on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree), whether the e-learning course provided adequate knowledge for the subsequent hands-on training. Additionally, they will assess their confidence in performing and interpreting the eFAST protocol. For the intervention group only, participants will also indicate whether they would have preferred in-person training instead of the teledidactic and whether they found the software/hardware easy to use.
Technical issues/usability | evaluation within 3 weeks after study completion
  Assessment whether participants in the intervention group encountered issues with the software or hardware used for the teledidactic training.
  Participants will indicate "yes" or "no" and, if they experienced issues, provide free-text explanations.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No